CLINICAL TRIAL: NCT02960737
Title: Dysphagia Evaluation After Stroke - a Randomized Controlled Trial of Oral Neuromuscular Training on Swallowing Dysfunction (DESIRE)
Brief Title: Dysphagia Evaluation After Stroke- Effect Oral Neuromuscular Training on Swallowing Dysfunction
Acronym: DESIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University Hospital, Umeå (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-319-31M
Record Dates: First submitted 2016-07-08; First posted 2016-11-10 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Dysphagia; Stroke
Keywords: Dysphagia; Stroke; Intervention; Oral neuromuscular training; Randomized control trial
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intensive training with oral neuromuscular training using an oral device (intervention group) and routine care with compensatory swallowing training under 3 months with start 12 (±3) weeks after stroke onset.
  Interventions: Device: Oral neuromuscular training using an oral device
- Control group (No Intervention): Routine care with compensatory swallowing training under 3 months with starting 12 (±3) weeks after stroke onset.

INTERVENTIONS:
Device: Oral neuromuscular training using an oral device — The oral device is used for 30 seconds, three times a day, before meals and implies new possibilities for training of the orofacial and pharyngeal muscles.
  Arms: Intervention group

SUMMARY:
The aim of this study is to investigate the effect of a specific rehabilitation program with an oral device used in stroke patients with persistent oral-and pharyngeal dysphagia.

DETAILED DESCRIPTION:
This study aims to investigate the effect of oral neuromuscular training in stroke patients with persistent oral- and pharyngeal dysphagia 12 (±3) weeks after stroke onset.

Interventional study with PROBE-design (prospective randomized open-label blinded evaluator). Consecutive patients with first-ever stroke without previously known dysphagia with persistent dysphagia (DOSS<6) at 3 months (12±3 weeks) post-stroke onset. Patients are eligible to participate if they are admitted to one of the following seven hospitals/centers in Sweden: Umeå University Hospital, Danderyds Hospital, Södersjukhuset, Skaraborg Hospital (Skövde), Helsingborg Hospital, Halland Hospital, Kungälv Hospital, Kalix Hospital, Skellefteå Hospital, and Ellenbogen in Malmö. Further centers will be recruited. Exclusion criteria: Unable/unwilling to give informed consent or to cooperate.

Randomization will be made web-based 1:1 by use of the developed REDCap system with stratification for center and aspiration (yes/no).

In total, 336 stroke patients (168 intervention group; 168 control group) with persistent dysphagia 12(±3) weeks after stroke onset will be included in the present study. The intervention group will be offered to undergo oral neuromuscular training alongside routine care with compensatory training for 3 months. The control group will only be offered routine care with compensatory training for 3 months.

The participants' status regarding swallowing function, nutritional status, quality of life related to swallowing, pneumonia, functional status including lip force, and death will be assessed before and after the completed intervention period, and 6 months post-intervention.

The primary endpoint will be analyzed using an ordinal regression (proportional odds) model, adjusting for baseline DOSS as well as for the stratifying variables center and aspiration.

The investigators hypothesize that swallowing intervention with oral neuromuscular training is more effective than routine care rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Persistent dysphagia 12(±3) weeks after STROKE.

Exclusion Criteria:

* Stroke patients with neurologic or psychiatric disorders or other diseases/conditions that can affect swallowing function.
* Unable to collaborate due to other serious diseases and/or to affected general condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Swallowing Function | At start compared with at end of treatment (after 3 months)
  Change in swallowing function measured by the Dysphagia Outcome Severity Scale (DOSS) using Fiberoptic endoscopic evaluation of swallowing (FEES)

SECONDARY OUTCOMES:
Swallowing function | At start and 6 months post-intervention
  Change in swallowing function measured by the Dysphagia Outcome Severity Scale (DOSS) using Fiberoptic endoscopic evaluation of swallowing (FEES)
Lip-force (LF) | At start, at end of treatment (after 3 months) and 6 months post-intervention
  Change in lip-force measured in newtons (N) with the Lip Force Meter LF100.
Swallowing Quality of Life Questionnaire (SWAL-QOL) | At start, at end of treatment (after 3 months) and 6 months post-intervention
  Change in quality of life related to swallowing measured by the SWAL-QOL questionnaire.
Nutritional status | At start, at end of treatment (after 3 months) and 6 months post-intervention
  Change in nutritional status measured with the Mini Nutritional Assessment (MNA).
Activity of daily living (ADL) | At start, at end of treatment (after 3 months) and 12-18 months post-intervention
  Change in activity of daily living (ADL) measured by Barthels Index (BI).
Global disability | At start, at end of treatment (after 3 months) and 6 months post-intervention
  Change in global disability measured with modified Rankin Scale (mRS)
Aspiration-pneumonia | At start, at end of treatment (after 3 months) and 6 months post-intervention
  Change in rate of aspiration-pneumonia based on the modified criteria by Centers for Disease Control and Prevention (CDC) for stroke-associated pneumonia
Death | At start, at end of treatment (after 3 months) and 6 months post-intervention
  Change in rate of death

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Hägglund, PhD/SLP, Principal Investigator — Umeå University
Locations (1):
- University Hospital of Umeå, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No